CLINICAL TRIAL: NCT05927974
Title: Investigating Dynamic Interactions in Distributed Cognitive Control Networks
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, J. Nicole Bentley, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300010350; UAB (Other: UAB)
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment; Dementia; ADD; Depression
Keywords: Cognitive tasks; Epilepsy; Intracranial EEG
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Depression; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICM Patients: Epillipsey Patients undergoing routine intracranial EEG monitoring for epilepsy.
  Interventions: Diagnostic Test: Passive testing; Diagnostic Test: Active testing

INTERVENTIONS:
Diagnostic Test: Passive testing — Passive testing includes baseline recordings or behavioral tasks without stimulation. Examples include language tasks, cognitive, and motor tasks. Passive testing typically takes 30-60 minutes and does not require presence of an epileptologist as the tasks are of minimal or no risk.
Diagnostic Test: Active testing — Active testing includes any study activity in which stimulation occurs. The most frequent paradigm consists of delivering small amounts of electrical stimulation through the implanted grid/strip/depth electrodes. This will be either continuous stimulation or patterned stimulation such as intermittent theta-burst . Stimulation will range between 1-8 mAmp. The duration of these pulses will last between 2-5 seconds.
  Subjects may be asked to rest quietly or to perform behavioral tasks during stimulation. Since there is a risk of evoking seizure activity with active testing, presence of an epileptologist is required. Active testing will only occur once the PI/staff has communicated with the epileptologist regarding safety, feasibility, and timing of active testing. Active testing will typically take 60-90 minutes and is only performed once patients are back on their anti-seizure medications.

SUMMARY:
The purpose of this study is to investigate the brain activity associated with cognitive tasks (thinking, reasoning, remembering) in order to understand how the brain works during certain tasks and to improve treatment for diseases like dementia and attention deficit disorders. Cognitive (thinking) impairment may include poor memory function, poor attention span, or psychiatric disorders (ex: ADD, depression). The investigators are interested in the brain activity related to these issues, and want to investigate changes in brain activity while we record activity from specific areas of the brain. These recordings are in addition to clinical (routine or standard of care) recordings being performed to monitor for seizures and do not impact the clinical care.

DETAILED DESCRIPTION:
Routine intracranial monitoring (ICM) surgery involves placement of several (10-20) electrodes into the brain through a small opening to a target structure. Participants have been deemed a surgical candidate for this procedure, and detailed discussion of the procedure will occur as part of the surgical consent. The Investigators may place sensors (stickers) to monitor participant's arm/hand movements and brain activity. Sensors may be placed on participant's scalp and/or arms and legs. The Investigators may place a device on participant's wrist or finger to measure position (accelerometer). The Investigators may perform voice recordings, eye movement tracking, and motion capture recordings to obtain measures of how stimulation affects speech and other movements. These are performed without any attachment of devices.

Cognitive tasks: Multiple cognitive tasks may be used and will be decided upon based on the clinical symptoms, exam, or comorbidities. These may include Go/No-go, Simon/Stroop task, Stop-signal task, language tasks, Tower of London, gambling task, maze navigation, choice-reaction time, delay tasks, and attention tasks.

Cortico-cortical evoked potentials and Patterned Stimulation: Stimulus pulses at precise time intervals and or various patterns will be delivered across adjacent electrode contacts at a series of electrode sites while simultaneously recording neural activity at other electrodes. This does not require any activity from participant.

Tasks will be administered via computer monitor positioned in front of the you. This will be connected to a recording computer. Participant will respond via keyboard, mouse, or response button.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for surgery based on multi-disciplinary consensus review
* Have a diagnosis of medically-refractory epilepsy
* A minimum of 18 years of age
* Willingness to participate in the paradigms described in the protocol

Exclusion Criteria:

* Inability to provide full and informed consent
* Age younger than 18
* Are not physically able to participate in study-related activities
* Major medical or surgical complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy undergo a routine surgery to implant electrodes into the brain for intracranial monitoring (ICM) to localize areas of the brain producing seizures.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-03-27 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Go/No-go | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Simon/Stroop task | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Stop-signal task | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Language task | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Tower of London | Post-op Day Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Gambling task | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Maze navigation | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Choice-reaction time | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Delay task | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Attention task | Post-op through study completion, an average of 7 days.
  Cognitive tasks given will be decided upon based on the clinical symptoms, exam, or comorbidities. Tasks will be administered via computer monitor positioned in front of the subject. This will be connected to a recording computer. Participants will respond via keyboard, mouse, or response button.
Cortico-cortical evoked potentials | Post-op through study completion, an average of 7 days.
  Stimulus pulses at precise time intervals will be delivered across adjacent electrode contacts at a series of electrode sites while simultaneously recording neural activity at other electrodes.
Patterned Stimulation | Post-op through study completion, an average of 7 days.
  Stimulus pulses at various patterns will be delivered across adjacent electrode contacts at a series of electrode sites while simultaneously recording neural activity at other electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica N Bentley, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No